CLINICAL TRIAL: NCT01628757
Title: Model Development and Prospective Validation to Predict the Response to Neoadjuvant Chemotherapy in Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ding Ma (Other)
Collaborators: Zhejiang University (Other); Shandong University (Other); Sun Yat-sen University (Other); Wuhan University (Other); Hubei Women and Children's Hospital (Unknown); Wuhan General Hospital of Guangzhou Military Command (Other); Xiangfan Central Hospital (Unknown); Wuhan Central Hospital (Other); Hubei University for nationalities (Unknown)
Responsible Party: Sponsor-Investigator, Ding Ma, Prof. of Dept. of O & G, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: GM2011-07-01; CERVca02/2002 (Other: HUST, ZJU, SDU，Sun Yat-sen University)
Record Dates: First submitted 2012-06-26; First posted 2012-06-27 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA from blood,TCT,pap smear,and hpv, as well as body fluid and tissues.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- neoadjuvant chemotherapy

SUMMARY:
Cervical cancer is one of the major health problems for chinese women. Besides surgery and radiotherapy, neoadjuvant chemotherapy has been proved to be an effective program by many studies.

However, not all patients respond well to neoadjuvant chemotherapy. Knowing the therapeutic effect of the neoadjuvant chemotherapy before receiving it can not only reduce the economic burden, but also more importantly save time to take more suitable treatments.

This study is undertaken to build a model combine both clinical and genetic factors to predict the effects of neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Cervical cancer has been one of the most commom malignant diseases among femails, and do a lot of harm to both young and older women, especially to the people in the undeveloped areas. Neoadjuvant chemotherapy has been investigated for treatment of cervical cancer patients since 1980s around the world（Sardi J, Di Paola G, Giaroli A, Sananes C, Burlando S and Rueda NG，1988；Mancuso S, Benedetti Panici P, Greggi S and Scambia G，1989.）. Clinicians found that neoadjuvant chemotherapy can help to diminish the tumor size,eliminate the distant metastasis; thus, patients can get the opportunity of surgery (Benedetti Panici P, Scambia G, Greggi S, Di Roberto P, Baiocchi G and Mancuso S，1988). As a result, women may have the chance to have their ovarian function preserved; and by plus surgery and post-surgery therapy, the women may also be able to be cured in the areas where sophisticated radiotherapy utilities are not availble.

As the development of science and techonology in chemotherapy for cervical cancer, the neoadjuvant therapy was also brought into China. And since 1990s, the investigation of neoadjuvant chemotherapy in China has been carried out in the teaching hospitals of China's leading famous universities in the developed aress. Strengthened by the prosperous economy of the countries, neoadjuvant chemotherapy began familar to China's Gyneclogists before the ending of the 20th century.

Since the beginning of the 21th century, that's in the early 2000s, neoadjuvant chemotherapy has been introduced as a new therapeutic therapy method. Neoadjuvant chemotherapy has also showed its own advantages (Chang TC, Lai CH, Hong JH, Hsueh S, Huang KG, Chou HH, Tseng CJ, Tsai CS, Chang JT, Lin CT, Chang HH, Chao PJ, Ng KK, Tang SG and Soong YK, 2000) and carried out in our hospitals, with the approvements of the institutions. Response both short-term and long-term response were evaluated. Clinical response, which is also known as early reponse, is also one of the short-term response, and has also been evaluated according to the response criterion. Patients' toxicity and long-term survival have also been recorded and evaluated. The treatment, as well as the study, was carried out in accordance with the approved guidelines. All eligible patients gave written informed consent before therapy. All protocols were approved by the ethical committees in the universities or the institutions, and updated with the renovated Declaration of Helsinki.

Since the middle stage or the late stage of 2000s, more clinicians have studied neoadjuvant chemotherapy in the top universities hospitals as well as our hospitals, and taken the chemotherapy regimens to the hospitals and institutions of theirs for the treatment of cervical cancer patients. Some of them have also taken part in the study with us.

And since the begining of the 2010s, more hospitals have taken part in the neoadjuvant study with us, and the number of the institutions have been updated with updation of protocols and ethical approvements. Patients who have fulfilled the inclusion criterion have been included with exclusion of disabled patients, such as Karnofsky Performance Status < 70，hepatic dysfunction, cardiac dysfunction and so on.

Although Concurrent Chemoradiotherapy has been treated as an standard treatment of cervical cancer (ref 4-6), neoadjuvant chemotherapy has also showed its own advantages (Chang TC, Lai CH, Hong JH, Hsueh S, Huang KG, Chou HH, Tseng CJ, Tsai CS, Chang JT, Lin CT, Chang HH, Chao PJ, Ng KK, Tang SG and Soong YK, 2000): it can facilitate premenopause women to have their ovarian function preserved in addition to the facility of radical surgery, some people have so good response that the tumor disappear completely after neosdjuvant chemotherapy. This may open an new window to young women who want to have their fertility (including uterus and ovaries) preserved. And the mechanism of chemotherapy-response and chemo-resistence in still need to be widely and deeply explored, which is also important for clinicians to understand the pathway of chemo-drugs' metablism and to avoid the toxic effect of the chemo-drugs.

ELIGIBILITY:
Inclusion Criteria:

* Untreated cervical cancer with FIGO stage Ib-IIIb
* Measurable lesions
* Possible to radical hysterectomy
* Age: 18 and older
* Karnofsky Performance Status≥ 70.
* WBC > 3,000/mm³, Hb > 9.0g/dl, Platelet > 100,000 /mm³, SGOT/SGPT < 60 IU/L, T-Bil < 1.5 mg/dL, Cr < 1.2 mg/dL, PaO2 > 80 torr, normal ECG
* Written informed consent

Exclusion Criteria:

* Previous history of cancer
* Patients with previous treatment
* Patients without information of clinical risk factors
* Patients who have active infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed Ib~ IIIb cervical carcinoma underwent Neoadjuvant Chemotherapy
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Primary Completion 2018-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The clinical and pathological response to neoadjuvant chemotherapy | 1 to 3 months
  including: ① clinical response（tumor size）, ②pathological response（<3 mm or not）, ③toxic response (degree) and so on.

SECONDARY OUTCOMES:
long-term response for patients undergoing neoadjuvant chemotherapy | up to 10 years to 20 years or more
  including ① DFS, ②OS, ③long-term complications，④secondary diseases, ⑤life quality, ⑥long-term toxic effects caused by the treatment and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China